CLINICAL TRIAL: NCT02945176
Title: A Prospective Open-label, Multicenter Clinical Investigation to Assess the Safety and Performance of ARGOS-IO System in Patients Undergoing Implantation of a Boston Keratoprosthesis (BKPro)
Brief Title: Safety and Performance Study of the ARGOS-IO System in Patients Undergoing Boston Keratoprosthesis Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Implandata Ophthalmic Products GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ARGOS-KP01; CIV-14-09-012725 (Registry Identifier: EUDAMED)
Record Dates: First submitted 2016-09-07; First posted 2016-10-26 (Estimated); Results first posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Graft vs Host Disease; Congenital Aniridia; Chemical Burns; Stevens-Johnson Syndrome; Congenital Glaucoma
Keywords: Boston Keratoprosthesis
MeSH Terms: conditions — Graft vs Host Disease; Aniridia; Burns, Chemical; Stevens-Johnson Syndrome; Hydrophthalmos

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ARGOS-IO system (Experimental): The ARGOS-IO system is a non-European Community (CE) marked investigational medical device composed of the implant and its accessories.
  Implant: ARGOS-IO pressure sensor implant for sulcus placement or transcleral fixation
  Accessories: MESOGRAPH reading device, Implant Injector
  Interventions: Device: ARGOS-IO system

INTERVENTIONS:
Device: ARGOS-IO system — This study will enroll a minimum of 10 and a maximum of 15 patients. It is anticipated to be large enough to provide an initial estimate of common safety events and assessment of performance. Any adverse event (AE), serious adverse event (SAE), ADE (adverse device event) and SADE (serious adverse device event) will be listed. Incidence will be estimated with a 95% confidence interval (Pearson-Clopper, two-sided). The Bland-Altman method will be used to assess the limits of agreement between the IOP measurements ARGOS-IO and surgical manometry. When appropriate, two-sided 95% confidence intervals, for these limits will be calculated accounting for repeated measurements based on the method proposed by Zou (2011). Other secondary performance endpoints will be analyzed by descriptive and explorative statistical methods.
  Other Names: ARGOS-IO pressure sensor implant

SUMMARY:
The ARGOS-IO pressure sensor is intended to be implanted in the human eye in combination with Boston Keratoprosthesis (BKPro) surgery and to remain in place indefinitely. It is intended to be used together with the hand-held Mesograph reading device to telemetrically measure the intraocular pressure (IOP) of patients with a BKPro.

The purpose of this study is to evaluate the safety and performance of the ARGOS-IO system in patients undergoing concomitant implantation of a BKPro and an ARGOS-IO sensor over the 12 month period beginning at implantation.

DETAILED DESCRIPTION:
(see above)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 18 and ≤ 80 years on the day of screening
2. Keratoprosthesis surgery indicated, defined as having a severely opaque and vascularized cornea AND either a verifiable history of two or more prior failed corneal transplant procedures or a medical condition such as alkali burns or autoimmune disease that makes the success of a traditional corneal transplant procedure unlikely. Potential study subjects will be solicited for participation in the clinical trial only after they have consented to the keratoprosthesis operation.
3. Axial length > 21 mm
4. Ability and willingness to attend all scheduled visits and comply with all study procedures

Exclusion Criteria:

1. Reasonable chance of success with traditional keratoplasty
2. Current retinal detachment
3. Connective tissue diseases
4. History or evidence of severe inflammatory eye diseases (i.e. uveitis, retinitis, scleritis) in one or both eyes within 6 months prior to ARGOS-IO implantation
5. History of ocular or periocular malignancy
6. History of extensive keloid formation
7. Any known intolerance or hypersensitivity to topical anesthetics, mydriatics, or silicone (component of the device)
8. Presence of another active medical eye implant and/or other active medical implants in the head/neck region
9. Signs of current infection, including fever and current treatment with antibiotics
10. Severe generalized disease that results in a life expectancy shorter than a year
11. Any clinical evidence that the investigator feels would place the subject at increased risk with the placement of the device
12. Currently pregnant or breastfeeding
13. Participation in any study involving an investigational drug or device within the past 30 days or ongoing participation in a study with an investigational drug or device
14. Intraoperative complication that would preclude implantation of the study device
15. Subject and/or an immediate family member is an employee of the investigational site directly affiliated with this study, the sponsor or the contract research organization.

Previous or concurrent enrollment of the contralateral eye in this clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-03; Primary Completion 2017-06-14 (Actual); Study Completion 2017-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Neuhann, Prof. MD, Principal Investigator — MVZ Prof. Neuhann
Locations (2):
- Germany (2):
  - Zentrum für Augenheilkunde der Universität zu Köln, Cologne
  - MVZ Prof. Neuhann, Munich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Telemetric Intraocular Pressure Monitoring after Boston Keratoprosthesis Surgery Using the Eyemate-IO Sensor: Dynamics in the First Year — https://doi.org/10.1016/j.ajo.2019.02.025

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from February 2015 to June 2016 in medical clinics.
Pre-assignment Details: 13 patients with an indication for a Boston Type I Keratoprosthesis (BI-KPro) were initially enrolled (13 = Safety Set (SS)*), 12 of whom successfully received the ARGOS-IO implant (12 = "ARGOS-IO system"-Group = Per-Protocol-Set (PPS)*) and were subjected to the follow-up visits. In one patient, the surgical preparation of the eye for implantation of the BI-KPro was so complex that the surgeon decided not to attempt implantation of the ARGOS-IO implant. *= as specified by the protocol
Groups:
- ARGOS-IO System: The ARGOS-IO Pressure sensor will be additionally implanted during local routine working procedures for Boston Keratoprosthesis (BKPro) surgery in patients undergoing implantation of a Boston Type I Keratoprosthesis (BI-KPro).
  ARGOS-IO system: Implantation of ARGOS-IO pressure sensor prior to fixation of the BI-KPro.
Period: Overall Study
Arm/Group | ARGOS-IO System
Started | 12 (13 patients with an indication for a Boston Type I Keratoprosthesis (BI-KPro) were initially enrolled (13 = Safety Set (SS), as specified by the protocol), 12 of whom successfully received the ARGOS-IO implant (12 = "ARGOS-IO system"-Group = Per-Protocol-Set (PPS), as specified by the protocol) and were subjected to the follow-up visits.)
Completed | 9
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- Safety Set: A total of 13 patients with an indication for BI-KPro implantation were initially enrolled in this open-label clinical investigation ("Safety Set"-Group), 12 of whom successfully received the ARGOS-IO implant. In one patient, the surgical preparation of the eye for implantation of the BI-KPro was so complex that the surgeon decided not to attempt implantation of the ARGOS-IO implant.
Arm/Group | Safety Set
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Germany | 13
Number of patients who successfully received the ARGOS-IO implant [Count of Participants; unit: Participants] | 12

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability: Number of Patients Experiencing a Device Related SAE (SADE)
Description: Number of patients experiencing a device-related SAE (SADE).
Time Frame: Assessed at visits from Day 0 [Implantation] through Week 52, final status at Week 52 reported.
Population: Safety: Number of Patients Experiencing a Device-related SAE (SADE)
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Set
Number analyzed (Participants) | 13
Participants
  Overall Number of Participants Analyzed | 13
  Number of Patients Experiencing a Device-related SAE (SADE) | 0

2. Primary Outcome: Performance: Performance of the ARGOS-IO System Compared to Manometry
Description: Consistency between manometric and telemetric IOP obtained by the ARGOS-IO system.
Time Frame: Assessed at visits Week 4, Week 16, Week 28 and Week 52, final status at Week 52 reported.
Population: IOP measurements with the ARGOS-IO system and by surgical manometry at given intervals (9 patients).
Measure: Count of Units; unit: Comparisons
Units Other Than Participants: Comparisons
Groups:
- ARGOS-IO System: The 12 patients whom successfully received the ARGOS-IO implant ("ARGOS-IO System"-Group), returned for 13 follow-up visits (V03-V15) consisting of comprehensive ophthalmic examinations as well as IOP measurements with the ARGOS-IO system and by finger palpation at all visits and manometric IOP measurements at defined intervals.
Arm/Group | ARGOS-IO System
Number analyzed (Participants) | 9
Number analyzed (Comparisons) | 24
Comparisons
  Consistency between manometric and telemetric IOP results with a deviation <10% in # of events | 9
  Consistency between manometric and telemetric IOP results with a deviation <20% in # of events | 14

3. Secondary Outcome: Safety and Tolerability: Incidence, Nature, Severity & Seriousness of Observed AEs/ADEs.
Description: Safety evaluation based on the incidence, nature, severity and seriousness of observed adverse events and adverse device events ("Frequency of Adverse Events").
  [Note that patients indicated for a BKPro surgery generally suffer from severe corneal disorders, reflected by the large number of AEs observed in this patient population.]
Time Frame: Assessed at visits from Day 0 [Implantation] through Week 52, final status at Week 52 reported.
Population: All available adverse events.
Measure: Number; unit: A(D)Es
Units Other Than Participants: A(D)Es
Groups:
- Safety Set: A total of 13 patients with an indication for BI-KPro implantation were initially enrolled in this open-label clinical investigation ("Safety Set"-Group), 12 of whom successfully received the ARGOS-IO implant (= IMD). In one patient, the surgical preparation of the eye for implantation of the BI-KPro was so complex that the surgeon decided not to attempt implantation of the ARGOS-IO implant.
Arm/Group | Safety Set
Number analyzed (Participants) | 13
Number analyzed (A(D)Es) | 168
A(D)Es
  Overall number of AEs/ADEs of which | 168
  AEs related to the medical procedure and/or | 116
  AEs unlikely related to the IMD and/or | 92
  AEs with no relation to the IMD and/or | 61
  AEs possibly related to the IMD | 15

4. Secondary Outcome: Performance: Correlation Between Finger Palpation and the ARGOS-IO System
Description: Correlation between IOP estimation obtained by finger palpation and the telemetric IOP by the ARGOS-IO system.
Time Frame: Assessed at visits from Day 1 through Week 52, final status at Week 52 reported.
Population: Intraocular pressure (IOP) estimation by finger palpation was grouped in 4 IOP categories: normal (A), soft/hypotonic (B), borderline (C) and hypertonic (D). Comparison measurements between finger palpation (IOP categories A/B/C/D) and telemetric IOP (in mmHg) by the ARGOS-IO system was carried out for all 12 patients. All available Finger Palpation estimates and ARGOS-IO measurements were analyzed (113 comparisons analyzed).
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: Comparisons
Arm/Group | ARGOS-IO System
Number analyzed (Participants) | 12
Number analyzed (Comparisons) | 113
mmHg
  Category A (normal): number analyzed (Participants) | 11
  Category A (normal): number analyzed (Comparisons) | 80
  Category A (normal) | 18.2 (6.1)
  Category B (soft/hypertonic): number analyzed (Participants) | 8
  Category B (soft/hypertonic): number analyzed (Comparisons) | 16
  Category B (soft/hypertonic) | 8.9 (2.8)
  Category C (borderline): number analyzed (Participants) | 5
  Category C (borderline): number analyzed (Comparisons) | 9
  Category C (borderline) | 22.4 (4.9)
  Category D (hypertonic): number analyzed (Participants) | 4
  Category D (hypertonic): number analyzed (Comparisons) | 8
  Category D (hypertonic) | 34.3 (11.0)

5. Secondary Outcome: Usability: User Acceptance at Home
Description: User acceptance of the ARGOS-IO system at home by means of evaluation of patient questionnaires on a score on a scale of 1 to 7 how strongly they agree to given statements (1 = totally disagree, 7 = totally agree). The score 7 represents a greater user acceptance.
Time Frame: Assessed at visit Week 52, final status at Week 52 reported.
Population: Each patient was asked to provide feedback on the user acceptance of the ARGOS-IO system at home. A total of 6 patients provided feedback via a structured questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARGOS-IO System
Number analyzed (Participants) | 6
score on a scale | 5.9 (3.0)

ADVERSE EVENTS:
Time Frame: Evaluation over 12 months follow-up period.
Description: SAE Definition
  That meets any of the following criteria of a serious adverse event:
  * Resulted in death, permanent damage or disability or a congenital anomaly
  * Was life threatening
  * Required hospitalization
Arm/Group | Safety Set
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 9/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Set (N=13)
Cystoid macular oedema (Eye disorders) | 2 (3)
Retinal detachment (Eye disorders) | 2 (2)
Retinopathy proliferative (Eye disorders) | 2 (2)
Corneal infiltrates (Eye disorders) | 1 (1)
Corneal perforation (Eye disorders) | 1 (1)
Hypotony of eye (Eye disorders) | 1 (1)
Iris adhesions (Eye disorders) | 1 (2)
Vitritis (Eye disorders) | 1 (1)
Complication associated with BI-KPro (General disorders) | 1 (1)
Transplant failure (Injury, poisoning and procedural complications) | 1 (1)
Intraocular pressure increased (Investigations) | 2 (2)
Device dislocation (Product Issues) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Corneal transplant (Surgical and medical procedures) | 2 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Set (N=13)
Eye pain (Eye disorders) | 6 (7)
Hypotony of eye (Eye disorders) | 5 (7)
Vitritis (Eye disorders) | 3 (4)
Keratitis (Eye disorders) | 2 (3)
Choroidal detachment (Eye disorders) | 2 (2)
Retinopathy proliferative (Eye disorders) | 2 (2)
Visual acuity reduced (Eye disorders) | 2 (2)
Procedural Pain (Injury, poisoning and procedural complications) | 3 (3)
Intraocular pressure increased (Investigations) | 6 (28)
Intraocular pressure decreased (Investigations) | 3 (4)
Retroprosthetic membrane (Product Issues) | 6 (7)
Device material opacification (BKPro and IOL) (Product Issues) | 3 (5)
Corneal sutures removal (Surgical and medical procedures) | 5 (8)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Cystoid macular edema (Eye disorders) | 1 (4)
Corneal epithelium defect (Eye disorders) | 1 (3)
Iris adhesion (Eye disorders) | 1 (2)
Ocular discomfort (Eye disorders) | 1 (2)
Trichiasis (Eye disorders) | 1 (2)
Anterior chamber cell (Eye disorders) | 1 (1)
Anterior chamber fibrin (Eye disorders) | 1 (1)
Blepharitis (Eye disorders) | 1 (1)
Choroidal haemorrhage (Eye disorders) | 1 (1)
Conjunctival disorder (Eye disorders) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 1 (1)
Corneal infiltrates (Eye disorders) | 1 (1)
Corneal neovascualrisation (Eye disorders) | 1 (1)
Erythema of eyelid (Eye disorders) | 1 (1)
Eye inflammation (Eye disorders) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1)
Keratic precipitates (Eye disorders) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1)
Lens disorder (Eye disorders) | 1 (1)
Pigment dispersion (Eye disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Retinal disorder (Eye disorders) | 1 (1)
Retinal haemorrhage (Eye disorders) | 1 (1)
Retinal scar (Eye disorders) | 1 (1)
Retinal tear (Eye disorders) | 1 (1)
Retinal thickening (Eye disorders) | 1 (1)
Subretinal fibrosis (Eye disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (1)
Vitreous opacities (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Atrophy of the donor cornea (General disorders) | 1 (1)
Subjectively worse impression (General disorders) | 1 (1)
Drug intolerance (General disorders) | 1 (1)
Bacterial disease carrier (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Hyphaema (Injury, poisoning and procedural complications) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Suture related complication (Injury, poisoning and procedural complications) | 1 (1)
Seidel Test positive (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/76/NCT02945176/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/76/NCT02945176/SAP_001.pdf